CLINICAL TRIAL: NCT00038246
Title: Phase I/II Study of Paclitaxel, Estramustine Phosphate and Thalidomide for Patients With Metastatic Androgen-Independent Prostate Carcinoma (AI-PCa)
Brief Title: Study of Paclitaxel, Estramustine Phosphate and Thalidomide for Patients With Metastatic Androgen-Independent Prostate Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-087; NCT00082693 (obsolete NCT alias)
Record Dates: First submitted 2002-05-29; First posted 2002-05-30 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estramustine; Thalidomide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalidomide, Taxol, Estramustine (Experimental): Thalidomide starting dose 200 mg by mouth every day once a week; Taxol 100 mg/m^2 by vein (IV) over 3 hours Day 3 and Day 10; Estramustine 140 mg by mouth three times a day on Days 1-5, 8-12.
  Interventions: Drug: Estramustine; Drug: Thalidomide; Drug: Paclitaxel (Taxol)

INTERVENTIONS:
Drug: Estramustine — 140 mg by mouth (po) three times a day on Days 1-5, 8-12
  Other Names: Emcyt; Estramustine Phosphate
Drug: Thalidomide — 200 mg by mouth every day once a week with dose escalation every week if no dose limiting toxicity.
  Other Names: Thalomid
Drug: Paclitaxel (Taxol) — 100 mg/m^2 by vein (IV) over 3 hours Day 3 and Day 10

SUMMARY:
The three study drugs (Thalidomide, Taxol, and Estramustine) used in this study are all chemotherapy drugs used in shrinking the cancer.

DETAILED DESCRIPTION:
1. Evaluate the maximum tolerated dose of oral daily thalidomide along with Paclitaxel (100 mg/m^2 as a 3-hour infusion weekly * 2, every 21 days) and oral estramustine phosphate (140 mg by mouth three times/day 5 days per week * 2 weeks, every 21 days) for patients with metastatic androgen-independent prostate carcinoma.
2. Evaluate the efficacy of this regimen for patients with metastatic Androgen-Independent Prostate Cancer who failed up to two prior non-paclitaxel containing chemotherapy regimens, as measured by:

   * 2A. The objective response rate and 'prostate-specific antigen (PSA) response rate' of the combination treatment in patients with AI-PCa progressing after chemotherapy.
   * 2B. Secondary endpoints: calculate time to disease progression, effect on performance status, analgesic consumption, and survival.
3. To evaluate the toxicity of the combination treatment in patients with metastatic AI-PCa progressing after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Histologic demonstration of adenocarcinoma of the prostate. Patients with variant histologies (ductal carcinoma, small cell carcinoma) are eligible only for the Phase I part of the trial, but are excluded from the Phase II. If no sample of the primary tumor was obtained, biopsy of a metastatic site is sufficient if the tissue stains positive for PSA. Some pathologic material must be available for review. Indicator need not be biopsy proven if the clinical presentation is characteristic.
* Androgen-Independent progression of prostate carcinoma, as shown by:

  1. Serum testosterone level of < 50 ng/dL or prior bilateral orchiectomy. Treatment to maintain castrate levels of testosterone (LHRH agonists) should continue, and
  2. Either symptomatic progression, or, if patient is asymptomatic, then a rising serum PSA in two occasions at least 1 week apart, with a minimum pre-treatment serum PSA of 5.
* Patients must be off anti-androgens, such as flutamide (Eulexin), bicalutamide (Casodex) or nilutamide (Nilandron). They must have no evidence of response at least 4 weeks (6 weeks for bicalutamide) since anti-androgen withdrawal (or progression at any time since anti-androgen withdrawal).
* Patients with nodal and/or visceral disease are eligible.
* Patients may have up to 2 prior chemotherapy regimens for prostate cancer, provided that more than 3 weeks have elapsed since the last treatment and patients have recovered from toxicity. Ketoconazole is considered chemotherapy. Prior Taxanes are allowed in both the Phase I and Phase II part of the trial. For the Phase II part of the study, patients must have progressed after >/= 1 and </= 2 prior chemotherapy regimens for prostate cancer (as neoadjuvant treatment or for metastatic disease).
* Up to one prior dose of Strontium-89 (Metastron) is allowed, if given more than 12 weeks prior to study entry. Patients may have had radiation therapy involving < 15% of the bone marrow (completed more than 3 weeks of initiation of the study).
* Previous treatment with PC-SPES, herbal / alternative medicines, anti-angiogenesis inhibitors, immunotherapy, or other non-androgen mediated pathways (such as epidermal growth factor receptor antagonists or farnesyl transferase inhibitors) is allowed, provided that there is unequivocal evidence of disease progression since completion of the therapy and more than 2 weeks have elapsed since last treatment.
* Patients must be at least 2 weeks from prior surgery.
* Adequate physiologic reserve as evidenced by:

  1. Life expectancy of at least 12 weeks
  2. Zubrod performance status of < 2.
  3. Age > 18 years old.
  4. No clinical history of heart disease and a normal elect electrocardiogram (EKG or ECG), OR an ejection fraction of at least 45% (by echocardiogram (ECHO), Multiple Gated Acquisition (MUGA) or ventriculography).
  5. serum glutamic pyruvic transaminase (SGOT/SGPT) and conjugated bilirubin less than twice the upper limit of normal.
  6. Serum creatinine < 2.0 mg/dl (or, if creatinine > 2 mg/dl, then a creatinine clearance of at least 35 ml/min (measured or estimated by the Cockcroft formula: CLcr= [(140-age) * weight (kg)] / [72 * serum creatinine (mg/dl)].
  7. Absolute neutrophil count (ANC)>1500/mm^3; Platelets >100,000/mm^3; hemoglobin > 9.0 gm/dl.

Exclusion Criteria:

* Patients with variant histologies (ductal or small cell carcinoma) are excluded from the phase II part of the trial (are eligible for the phase I part).
* Patients with no prior chemotherapy for prostate cancer are excluded from the phase II part of the study.
* Patients with central nervous system (CNS) metastases or serious medical illnesses, active or uncontrolled infections, significant psychiatric disorders that preclude giving informed consent, patients with NCI grade > 2 peripheral neuropathy or patients with a history of another malignancy (except from superficial bladder cancer or basal cell carcinoma of the skin) within 5 years prior to study entry are excluded from the trial.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2000-10; Primary Completion 2004-02 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) Thalidomide | 21 day cycles
  MTD defined by Continuous reassessment method.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. Logothetis, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org